CLINICAL TRIAL: NCT05570240
Title: The Relationship Between Chronic OA Pain and Cognition Deficits in OA Patients.
Status: Completed | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chun-Hsien Wen, Physician, Kaohsiung Veterans General Hospital.
Other Study IDs: VGHKS19-CT2-21
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Knee Osteoarthritis; Neuroinflammatory Response
Keywords: Chronic pain; Knee osteoarthritis; Cognitive deficits
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OA group: Knee osteoarthritis patients who were scheduled to receive elective total knee replacement surgery which need spinal anesthesia.
- Control group: Control group patients were scheduled to receive elective general surgery or urological surgery with spinal anesthesia.

SUMMARY:
The goal of this observational study is to learn about the association between pain characteristics and cognitive functions in chronic knee osteoarthritis. The main questions it aims to answer are:

1. If pain characteristics affect cognitive functions in severe knee OA patients?
2. If concentration of neuroinflammation mediators were raised in severe knee OA patients with comparing with control group participants?

Participants will receive pain and cognition questionnaire before surgery and their blood and CSF will be collected for further analysis of neuroinflammation mediators.

DETAILED DESCRIPTION:
In the previous studies, which revealed that because neural systems involved in cognition and pain processing are closely linked, they may affect with each other. In addition to sensory symptoms, cognitive functioning is thought to be affected in chronic pain patients. Pain uses cognitive resources, alters neural plasticity and affects expression and activity of a variety of chemical and cellular neuromediators. There are several brain regions such as amygdala and hippocampus which are most commonly activated during pain processing.Osteoarthritis (OA) of the knee is one of the leading causes of disability among noninstitutionalized elderly adults. One population-based study revealed that osteoarthritis increases the risk of cognitive deficits diseases such as dementia. However the possible mechanism had not be elucidated. Recent study revealed that OA-induced hyperalgesia was associated with increased nerve growth factor (NGF)/tropomycin receptor kinase A (TrkA) signaling. NGF activation of extracellular signal-regulated kinase (ERK)/ mitogen-activated protein kinase (MAPK) may play a role in centralization of OA pain. Otherwise NGF has also been shown to produce a dramatic upregulation of brain-derived neurotrophic factor (BDNF) in trkA-expressing dorsal root ganglion (DRG) cells, and there is now growing evidence that BDNF may serve as a central regulator of excitability and is a neuromodulate or of central pain processing. On the other hand, in previous studies they showed that BDNF plays a critical role in synaptic plasticity, memory processes and storage of long-term memory. The BDNF/tropomycin receptor kinase B (TrkB) system in the hippocampus plays a crucial role not only in the memory acquisition, but also in the retention and / or recall of spatial memory.

Besides ongoing pain in chronic knee OA is characterized by increased brain activity in limbic-affective regions thus providing novel evidence for a strong emotional component of arthritis pain. There are feedback loops exist between pain, emotion and cognition. How is the role of BDNF in such loop? The objective of the study was the evaluation of association between pain characteristics and cognitive functions in severe knee OA patients. Besides, we will try to explore the possible mechanisms by which chronic OA like pain develops to cognitive deficits in animal models. The relationship between BDNF levels in body fluids (serum and CSF) and pain characteristics and cognitive function was also evaluated in the whole sample.

ELIGIBILITY:
Inclusion Criteria:

* OA patients who were scheduled to receive elective surgery which need spinal anesthesia.
* Age is more than 20 years old.
* American Society of Anesthesiologists (ASA) class I-III.

Exclusion Criteria:

* Unwilling to participate.
* Age is lesser than 20 years old.
* Autoimmune diseases.
* Previous knee injury or infection history.
* Brain region disease ex: stroke or brain tumor...etc.
* Mild cognitive impairment, dementia or other neurodegenerative diseases.
* Cancer.
* With other chronic pain.

Ages: 20 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with chronic knee osteoarthritis pain who will receive total knee replacement surgery. They have no other chronic pain except chronic knee pain. Furthermore they did not have any cerebral diseases such as stroke or brain tumor.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster universities Osteoarthritis Index (WOMAC) | The WOMAC questionnaire were measured on the day before their surgery.
  The WOMAC questionnaire has been used to assess subjects with OA of the hip or knee and consists of 24 items divided into 3 subscales: self-perception of pain (5 items), joint stiffness (2 items), and functional performance (17 items) during the previous 72 h.
The cognitive abilities screening instrument (CASI) | The CASI questionnaire were measured on the day before their surgery.
  The CASI has been commonly used in dementia research and clinical practice to evaluate a subject's cognitive abilities.
Glia mediators of neuroinflammation | All blood and CSF samples were obtained before spinal anesthesia.
  Glia mediators of neuroinflammation include interleukin-1β (IL-1β), interleukin-6 (IL-6), tumor necrosis factor α (TNF α), BDNF and fractalkine.

SECONDARY OUTCOMES:
The geriatric depression scale (GDS-15) | The GDS-15 questionnaire were measured on the day before their surgery.
  The GDS-15 was used for evaluation of emotion especially for participant of age > 65. years old.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Hsien Wen, Physician, Principal Investigator — Kaohsiung Veterans General Hospital.; Chen-Hsiu Chen, Physician, Study Director — Kaohsiung Veterans General Hospital.; Yuan-Yi Chia, Director, Study Director — Kaohsiung Veterans General Hospital.; Chih-Chi Tsai, RA, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hopital, Kaohsiung City, Zuoying Dist, Taiwan

REFERENCES:
- [Result] Zhang Y, Jordan JM. Epidemiology of osteoarthritis. Clin Geriatr Med. 2010 Aug;26(3):355-69. doi: 10.1016/j.cger.2010.03.001. PMID 20699159
- [Result] Kyrkanides S, Tallents RH, Miller JN, Olschowka ME, Johnson R, Yang M, Olschowka JA, Brouxhon SM, O'Banion MK. Osteoarthritis accelerates and exacerbates Alzheimer's disease pathology in mice. J Neuroinflammation. 2011 Sep 7;8:112. doi: 10.1186/1742-2094-8-112. PMID 21899735
- [Result] Huang SW, Wang WT, Chou LC, Liao CD, Liou TH, Lin HW. Osteoarthritis increases the risk of dementia: a nationwide cohort study in Taiwan. Sci Rep. 2015 May 18;5:10145. doi: 10.1038/srep10145. PMID 25984812
- [Result] Li X, Tong Q, Gao J, Liu C; Alzheimer's Disease Neuroimaging Initiative; Liu Y. Osteoarthritis Was Associated With a Faster Decline in Hippocampal Volumes in Cognitively Normal Older People. Front Aging Neurosci. 2020 Aug 14;12:190. doi: 10.3389/fnagi.2020.00190. eCollection 2020. PMID 32922280
- [Result] Wu L, Wang X, Ye Y, Liu C. Association of Osteoarthritis With Changes in Structural Neuroimaging Markers Over Time Among Non-demented Older Adults. Front Aging Neurosci. 2021 Aug 10;13:664443. doi: 10.3389/fnagi.2021.664443. eCollection 2021. PMID 34447303
- [Result] Clark AK, Malcangio M. Fractalkine/CX3CR1 signaling during neuropathic pain. Front Cell Neurosci. 2014 May 7;8:121. doi: 10.3389/fncel.2014.00121. eCollection 2014. PMID 24847207
- [Result] Grace PM, Hutchinson MR, Maier SF, Watkins LR. Pathological pain and the neuroimmune interface. Nat Rev Immunol. 2014 Apr;14(4):217-31. doi: 10.1038/nri3621. Epub 2014 Feb 28. PMID 24577438
- [Result] Montague K, Malcangio M. The therapeutic potential of targeting chemokine signalling in the treatment of chronic pain. J Neurochem. 2017 May;141(4):520-531. doi: 10.1111/jnc.13927. Epub 2017 Feb 24. PMID 27973687
- [Result] Subbarayan MS, Joly-Amado A, Bickford PC, Nash KR. CX3CL1/CX3CR1 signaling targets for the treatment of neurodegenerative diseases. Pharmacol Ther. 2022 Mar;231:107989. doi: 10.1016/j.pharmthera.2021.107989. Epub 2021 Sep 4. PMID 34492237
- [Result] Cappoli N, Tabolacci E, Aceto P, Dello Russo C. The emerging role of the BDNF-TrkB signaling pathway in the modulation of pain perception. J Neuroimmunol. 2020 Dec 15;349:577406. doi: 10.1016/j.jneuroim.2020.577406. Epub 2020 Sep 24. PMID 33002723
- [Result] Malfait AM, Miller RE, Block JA. Targeting neurotrophic factors: Novel approaches to musculoskeletal pain. Pharmacol Ther. 2020 Jul;211:107553. doi: 10.1016/j.pharmthera.2020.107553. Epub 2020 Apr 18. PMID 32311372
- [Result] Tang J, Bair M, Descalzi G. Reactive Astrocytes: Critical Players in the Development of Chronic Pain. Front Psychiatry. 2021 May 28;12:682056. doi: 10.3389/fpsyt.2021.682056. eCollection 2021. PMID 34122194

DOCUMENTS (1):
  • Study Protocol (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT05570240/Prot_000.pdf